CLINICAL TRIAL: NCT00381849
Title: Cystone for Treatment of Nephrolithiasis
Brief Title: Use of an Herbal Preparation to Prevent and Dissolve Kidney Stones
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Himalaya Herbal Healthcare (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Stephen B. Erickson, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2115-05; P50DK083007 (NIH)
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Results first posted 2012-08-06 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Cystinuria; Nephrolithiasis, Calcium Oxalate
Keywords: Cystone; Uricare; Computerized tomography; Kidney calculi; Supersaturation; Nephrolithiasis; Quantitative CT
MeSH Terms: conditions — Cystinuria; Nephrolithiasis, Calcium Oxalate; Kidney Calculi; Nephrolithiasis | interventions — cystone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cystone then sugar pill (Active Comparator): Subject will take Cystone for 6 weeks, then have a 1 week wash out period followed by the sugar pill for another 6 weeks
  Interventions: Drug: Cystone; Drug: Sugar Pill (Placebo)
- Sugar pill then Cystone (Placebo Comparator): Subject will take sugar pill for 6 weeks, then a 1 week wash out followed by the Cystone for another 6 weeks
  Interventions: Drug: Cystone; Drug: Sugar Pill (Placebo)
- Open-label Cystone (Experimental): All subjects will receive Cystone for 46 weeks in the open-label period.
  Interventions: Drug: Cystone

INTERVENTIONS:
Drug: Cystone — Participants will take 2 pills, 2 times a day.
  Each tablet of Cystone contains:
  Shilapushpha (Didymocarpus pedicellata) 130 mg, Pasanabheda (Saxifraga ligulata Syn. Bergenia ligulata/cilata) 98 mg, Indian madder/ Manjishtha (Rubia cordifolia) 32 mg, Umbrella's edge/ Nagarmusta (Cyperus scariosus) 32 mg, Prickly chaff flower/ Apamarga (Achyranthes aspera) 32 mg, Sedge/ Gojiha (Onosma bracteatum) 32 mg, Purple fleabane/ Sahadeve (Veronoia Cinerea) 32 mg, Lime silicate calx/ Hajrul yahood Bhasma/ Badrashma bhasma) 32 mg, Shilajit 26 mg.
  Other Names: Uricare
Drug: Sugar Pill (Placebo) — Participants will take 2 pills, 2 times a day for 6 weeks.
  Arms: Cystone then sugar pill; Sugar pill then Cystone

SUMMARY:
We will investigate the safety and effectiveness of a mixture of 9 east Indian herbs known as Cystone regarding their ability to dissolve existing kidney stones and prevent formation of new ones. Cystine and calcium stone formers will be recruited for a 59 week trial. The first phase of the study will be two 6 weeks periods during which each subject will receive Cystone or placebo in random order (with a one-week wash out between 6 week treatment periods). The remaining 46 weeks, each subject will receive Cystone. End points are changes in urinary chemistries and stone burden by Computerized Tomography (CT) scanning.

DETAILED DESCRIPTION:
Cystone will be used in proven cystine and calcium stone forming adults who are not pregnant. Subjects must have a measurable stone by CT. The first phase is a double blind, randomized, placebo controlled cross-over of Cystone and placebo for 6 weeks each separated by a 1 week washout. Entry, 6 and 12 week 24 hour urine supersaturations or cystine, pH and sodium determinations will be collected. Then all patients enter an open label phase of 46 weeks, ensuring a 52-week total exposure to Cystone during the 59 week study. Baseline and 1 year stone quantification CT scans will be performed. End points will be changes in urine chemistry/supersaturation and stone burden. Stone burden was measured by CT, quantitatively for stone density and volume. All CT images were also reviewed in a blinded fashion by a radiologist to score each kidney as increased, no change or decreased stone burden.

Statistics and Randomization: Randomization was accomplished using a table provided by the department of statistics to the study coordinator who was blinded as to whether the patients received placebo or Cystone®. Biochemical and supersaturation results were analyzed via a matched pair analysis using the JMP software package (SAS Instituted, Inc.); P values < 0.05 were deemed significant.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent In the cystine arm, all patients will have the diagnosis of cystinuria, made on the basis of a 24-hour urine cystine containing more than 1500 umol of cystine, or a stone compositional analysis of cystine
* Presence of an existing cystine stone in one or both kidneys In the calcium arm, all patients will have a history of a calcium stone as determined by laboratory analysis.
* Medically effective birth control if fertile female
* Able to comply with protocol

Exclusion Criteria:

* Pregnant
* Subjects under age 18 years
* Obstructing stones
* Urinary Tract Infection that cannot be cleared with single course of antibiotic
* Subjects who decline to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2009-09 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B. Erickson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Abdollahiasl A, Kebriaeezadeh A, Nikfar S, Farshchi A, Ghiasi G, Abdollahi M. Patterns of antibiotic consumption in Iran during 2000-2009. Int J Antimicrob Agents. 2011 May;37(5):489-90. doi: 10.1016/j.ijantimicag.2011.01.022. Epub 2011 Mar 17. No abstract available. PMID 21419606
- [Result] Erickson SB, Vrtiska TJ, Canzanello VJ, Lieske JC. Cystone(R) for 1 year did not change urine chemistry or decrease stone burden in cystine stone formers. Urol Res. 2011 Jun;39(3):197-203. doi: 10.1007/s00240-010-0334-x. Epub 2010 Dec 16. PMID 21161651

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with recurring and analytically confirmed kidney stones were recruited from the Mayo Stone Clinic in Rochester, MN.
Groups:
- Calcium Stone Subjects: Subjects with confirmed calcium kidney stone(s)
- Cystine Stone Subjects: Subjects with confirmed cystine kidney stone(s)
Period: First Intervention
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Wash Out
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Open-label
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Urine Supersaturation of Calcium Oxalate (CaOx)
Description: Urine is often supersaturated, which favors precipitation of crystalline phases such as calcium oxalate. However, crystals do not always form in supersaturated urine because supersaturation is balanced by crystallization inhibitors that are also present. Supersaturation is calculated by measuring the concentration of all the ions that can interact. Once these concentrations are known, a computer program can calculate the theoretical supersaturation with respect to the important crystalline phases, eg, calcium oxalate.
Time Frame: baseline, after 6 weeks treatment on placebo, after 6 weeks treatment on cystone, at end of 46 weeks of open label cystone treatment
Population: CaOx was not analyzed for the Cystine Stone subjects.
Measure: Mean (Standard Deviation); unit: KJoules/mol
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Number analyzed (Participants) | 10 | 0
KJoules/mol
  CaOx at Baseline | 1.83 (0.28) |
  CaOx after placebo (6 wks) | 1.83 (0.42) |
  CaOx after Cystone (6 wks) | 1.87 (0.43) |
  CaOx at end of Cystone (46 weeks) | 1.78 (0.47) |
Statistical Analysis 1: Comparison: Calcium Stone Subjects; Paired t test for supersaturation of CaOx between baseline and after 6 weeks' treatment on placebo; Test type: Superiority or Other; p = 0.32, t-test, 1 sided
Statistical Analysis 2: Comparison: Calcium Stone Subjects; Paired t test for supersaturation of CaOx between baseline and after 6 weeks' treatment on cystone; Test type: Superiority or Other; p = 0.23, t-test, 1 sided
Statistical Analysis 3: Comparison: Calcium Stone Subjects; Paired t test for supersaturation of CaOx between six weeks' treatment on cystone and 6 weeks' treatment on placebo; Test type: Superiority or Other; p = 0.41, t-test, 1 sided
Statistical Analysis 4: Comparison: Calcium Stone Subjects; Paired t test for supersaturation of CaOx between baseline and after 46 weeks' treatment on cystone; Test type: Superiority or Other; p = 0.32, t-test, 1 sided

2. Primary Outcome: 24 Hour Urine Supersaturation of Calcium Phosphate (Brushite)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Brushite was not analyzed for the Cystine Stone subjects.
Measure: Mean (Standard Deviation); unit: KJoules/mol
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Number analyzed (Participants) | 10 | 0
KJoules/mol
  Brushite at Baseline | 0.35 (1.04) |
  Brushite after placebo (6 wks) | 0.73 (0.83) |
  Brushite after Cystone (6 wks) | 0.38 (0.98) |
  Brushite at end of Cystone (46 weeks) | 0.09 (1.29) |
Statistical Analysis 1: Comparison: Calcium Stone Subjects; Paired t test for supersaturation of Brushite between baseline and after 6 weeks' treatment on placebo; Test type: Superiority or Other; p = 0.49, t-test, 1 sided
Statistical Analysis 2: Comparison: Calcium Stone Subjects; Paired t test for supersaturation of Brushite between baseline and after 6 weeks' treatment on cystone; Test type: Superiority or Other; p = 0.64, t-test, 1 sided
Statistical Analysis 3: Comparison: Calcium Stone Subjects; Paired t test for supersaturation of Brushite between six weeks' treatment on cystone and 6 weeks' treatment on placebo; Test type: Superiority or Other; p = 0.72, t-test, 1 sided
Statistical Analysis 4: Comparison: Calcium Stone Subjects; Paired t test for supersaturation of Brushite between baseline and after 46 weeks' treatment on cystone; Test type: Superiority or Other; p = 0.84, t-test, 1 sided

3. Primary Outcome: 24 Hour Urine Supersaturation of Calcium Phosphate (Hydroxyapatite)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Hydroxyapatite was not analyzed for the Cystine Stone subjects.
Measure: Mean (Standard Deviation); unit: KJoules/mol
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Number analyzed (Participants) | 10 | 0
KJoules/mol
  Hydroxyapatite at Baseline | 4.25 (2.02) |
  Hydroxyapatite after placebo (6 wks) | 5.03 (1.23) |
  Hydroxyapatite after Cystone (6 wks) | 4.65 (1.86) |
  Hydroxyapatite at end of Cystone (46 weeks) | 4.09 (2.06) |

4. Secondary Outcome: Change in Stone Burden as Assessed by Radiologist at One Year
Description: Stone burden will be quantitated using the stone quantification protocol currently available at Mayo that quantitates kidney stones both by volume and by density measured in Agatston units.
Time Frame: Baseline, approximately 52 weeks after baseline
Population: One subject in the Calcium group was excluded from the CT analysis because of bilateral stone removal surgery during the study.
Measure: Number; unit: Kidneys
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Number analyzed (Participants) | 9 | 9
Kidneys
  Right kidney no change in stone burden | 6 | 7
  Right kidney stone burden increased | 2 | 2
  Right kidney stone burden decreased | 1 | 0
  Left kidney no change in stone burden | 2 | 2
  Left kidney stone burden increased | 6 | 5
  Left kidney stone burden decreased | 1 | 2

5. Primary Outcome: 24 Hour Urinary Cystine Excretion
Time Frame: as for outcome 1
Population: Cystine excretion was not applicable to the Calcium Stone subjects.
Measure: Mean (Standard Deviation); unit: mcmol/24 hours
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Number analyzed (Participants) | 0 | 10
mcmol/24 hours
  Cystine at Baseline |  | 2770 (947)
  Cystine after placebo (6 wks) |  | 3183 (1898)
  Cystine after Cystone (6 wks) |  | 2948 (2021)
  Cystine at end of Cystone (46 weeks) |  | 4140 (2398)
Statistical Analysis 1: Comparison: Cystine Stone Subjects; Paired t test for urinary cystine between baseline and after 6 weeks' treatment on placebo; Test type: Superiority or Other; p = 0.69, t-test, 1 sided
Statistical Analysis 2: Comparison: Cystine Stone Subjects; Paired t test for urinary cystine between baseline and after 6 weeks' treatment on cystone; Test type: Superiority or Other; p = 0.25, t-test, 1 sided
Statistical Analysis 3: Comparison: Cystine Stone Subjects; Paired t test for urinary cystine between six weeks' treatment on cystone and 6 weeks' treatment on placebo; Test type: Superiority or Other; p = 0.15, t-test, 1 sided
Statistical Analysis 4: Comparison: Cystine Stone Subjects; Paired t test for urinary cystine between baseline and after 46 weeks' treatment on cystone; Test type: Superiority or Other; p = 0.20, t-test, 1 sided

6. Primary Outcome: Stone Density as Measured by Agatston Score Via Computerized Tomography
Description: Agatston results are a measure of calcium typically used for measuring coronary artery calcification.
Time Frame: Baseline, approximately 52 weeks after baseline
Population: One subject was excluded from CT analysis because of bilateral stone removal surgery during the study
Measure: Mean (Standard Deviation); unit: Agatston Score
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Number analyzed (Participants) | 9 | 10
Agatston Score
  Baseline Right Kidney Agatston Score | 49.75 (60.24) | 2,107 (4,417)
  52 week Right Kidney Agatston Score | 56.13 (74.23) | 2,183 (4,157)
  Baseline Left Kidney Agatston Score | 166.13 (143.16) | 383 (560)
  52 week Left Kidney Agatston Score | 247.71 (371.46) | 1,801 (2,741)
Statistical Analysis 1: Comparison: Calcium Stone Subjects; Right Kidney Stone Density; P-value comparing one year to baseline; Test type: Superiority or Other; p = 0.85, t-test, 2 sided
Statistical Analysis 2: Comparison: Calcium Stone Subjects; Left Kidney Stone Density; P-value comparing one year to baseline; Test type: Superiority or Other; p = 0.63, t-test, 2 sided
Statistical Analysis 3: Comparison: Cystine Stone Subjects; Right Kidney Stone Density; P-value comparing one year to baseline; Test type: Superiority or Other; p = 0.97, t-test, 2 sided
Statistical Analysis 4: Comparison: Cystine Stone Subjects; Left Kidney Stone Density; P-value comparing one year to baseline; Test type: Superiority or Other; p = 0.15, t-test, 2 sided

7. Primary Outcome: Volume of Kidney Stones as Measured on Computerized Tomography
Description: Measurement of kidney stone volume in cubic millimeters.
Time Frame: Baseline, approximately 52 weeks after baseline
Population: One subject was excluded from CT analysis because of bilateral stone removal surgery during the study.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Number analyzed (Participants) | 9 | 10
mm^3
  Baseline Right Kidney Stone Volume | 45.5 (52.03) | 1,602 (3,335)
  52 Week Right Kidney Stone Volume | 52.75 (66.44) | 1,677 (3,139)
  Baseline Left Kidney Stone Volume | 141.25 (198.98) | 301 (422)
  52 Week Left Kidney Stone Volume | 174.25 (265.73) | 2,064 (688)
Statistical Analysis 1: Comparison: Calcium Stone Subjects; Right Kidney Stone Volume; P-value comparing one year to baseline; Test type: Superiority or Other; p = 0.81, t-test, 2 sided
Statistical Analysis 2: Comparison: Calcium Stone Subjects; Left Kidney Stone Volume; P-value comparing one year to baseline; Test type: Superiority or Other; p = 0.78, t-test, 2 sided
Statistical Analysis 3: Comparison: Cystine Stone Subjects; Right Kidney Stone Volume; P-value comparing one year to baseline; Test type: Superiority or Other; p = 0.96, t-test, 2 sided
Statistical Analysis 4: Comparison: Cystine Stone Subjects; Left Kidney Stone Volume; P-value comparing one year to baseline; Test type: Superiority or Other; p = 0.13, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Description: Subject self reported any adverse effects.
Arm/Group | Calcium Stone Subjects | Cystine Stone Subjects
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
There were no serious adverse events and no adverse events. Power of the study was diminished by failure of patients to return all required 24 hour urine samples. The botanical authenticity of Cystone was not documented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No